CLINICAL TRIAL: NCT03343587
Title: A Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY3375880 in Healthy Subjects
Brief Title: A Study of LY3375880 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16833; I9N-MC-FCAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3375880 Single Dose (Experimental): Single dose of LY3375880 administered IV or SC
  Interventions: Drug: LY3375880 IV; Drug: LY3375880 SC
- Placebo Single Dose (Placebo Comparator): Single dose of placebo administered IV or SC
  Interventions: Drug: Placebo IV; Drug: Placebo SC
- LY3375880 Multiple Dose (Experimental): Multiple doses of LY3375880 administered IV or SC
  Interventions: Drug: LY3375880 IV; Drug: LY3375880 SC
- Placebo Multiple Dose (Placebo Comparator): Multiple doses of placebo administered IV or SC
  Interventions: Drug: Placebo IV; Drug: Placebo SC

INTERVENTIONS:
Drug: LY3375880 IV — administered IV
  Arms: LY3375880 Multiple Dose; LY3375880 Single Dose
Drug: LY3375880 SC — administered SC
  Arms: LY3375880 Multiple Dose; LY3375880 Single Dose
Drug: Placebo IV — administered IV
  Arms: Placebo Multiple Dose; Placebo Single Dose
Drug: Placebo SC — administered SC
  Arms: Placebo Multiple Dose; Placebo Single Dose

SUMMARY:
The purpose of this study is to evaluate how well LY3375880 (study drug) is tolerated in healthy participants and what side effects may occur. The study drug will be administered either subcutaneously (SC) under the skin or intravenously (IV) into a vein in the arm.

This is a two-part study. Participants will enroll in only one part. Part one will last about 16 weeks including screening and follow-up. This part will include 2 nights at the study site. Part two will last about 20 weeks including screening and follow-up. This part will include 2 nights at the study site for each dose.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* Have a body mass index of 18.0 to 32.0 kilograms per meter squared (kg/m²) inclusive
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* Have known allergies to LY3375880, related compounds or any components of the formulation, or history of significant atopy
* Are women who are of childbearing potential or who are lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Pre-dose to 3 months after administration of study drug
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3375880 | Pre-dose to 3 months after administration of study drug
  PK: Cmax of LY3375880
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3375880 | Pre-dose to 3 months after administration of study drug
  PK: AUC of LY3375880

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Parexel Early Phase Unit at Glendale, Glendale, California, United States